CLINICAL TRIAL: NCT04835285
Title: Clinical Study of MRI Assessment of Iron in the Myocardium, Liver, Pancreas and Pituitary Gland in Patients With High Transfusion Dependence on the Packed Red Blood Cells
Brief Title: MRI T2* Mapping of Myocardium, Liver, Pancreas and Pituitary Gland
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCPHOI-2019-09
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Iron Overload
Keywords: Iron; T2* mapping; MRI relaxometry; transfusion
MeSH Terms: conditions — Iron Overload

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Npf. — 3T MRI and 1,5 T MRI scanners. For myocardium, pancreas and pituitary gland iron overload

SUMMARY:
All patients were investigated using a 3T MRI and 1,5 T MRI scanners. For myocardium, pancreas and pituitary gland iron overload quantification in children we have used special sequences for T2*-mapping.

Miocardium, pancreas and pituitary gland T2* relaxometry maps were calculated automatically by commertial application ReportCARD Functool (GE Healthcare) and integrated Philips T2* maps. Then for selected ROI T2* data acquisition in milisecond [ms] were performed and calculated automatically.

DETAILED DESCRIPTION:
All patients were investigated using a 3T MRI scanner (Philips Achieva) and 1,5 T MRI scanner (GE Signa) with 8-channel surface coil for body scanning. For myocardium, pancreas and pituitary gland iron overload quantification in children we have used special sequences for T2*-mapping based on fast gradient echo sequences - multi-phase fast gradient echo and ultrashort gradient echo (uTE) in axial and coronary plane. For breath-hold acquisition due to failure of communication and invariable behavior some children received anaesthetic support with mechanical ventilation. Miocardium, pancreas and pituitary gland T2* relaxometry maps were calculated automatically by commertial application ReportCARD Functool (GE Healthcare) and integrated Philips T2* maps.

The placement of region of interest (ROI) in target organ were performed by following criterion: for the myocardium - in the interventricular septum in short axis plane; for the pancreas - in corpus in axial plane; for the pituitary gland - in adenohypophysis; for all organs the area of large and small blood vessels, which can introduce distortions of the obtained results were excluded. Then for selected ROI T2* data acquisition in milisecond [ms] were performed and calculated automatically by approximating the attenuation curve with the highest likelihood method.

ELIGIBILITY:
Inclusion criteria:

1. Age under 25 y.o.;
2. A history of transfusion-dependent anemia of various origins.
3. indications for the appointment of chelation therapy

Non-inclusion criteria:

1. Age over 25 y.o.
2. The number of RBC transfusions previously received by the patient is less than 10

Exclusion criteria:

1. Absolute contraindications to magnetic resonance imaging (pacemaker, ferromagnetic implants, etc.);
2. Refusal to sign the informed consent.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 152 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-01-21 (Estimated); Study Completion 2023-01-21 (Estimated)

PRIMARY OUTCOMES:
Compare and contrast T2* values in pancreas, myocardium, and pituitary gland in patients with transfusion-dependent anemia using 1.5T and 3T MRI scanner. | Initially, after one month of chelation therapy
Compare and contrast T2* values in pancreas, myocardium, and pituitary gland in patients with transfusion-dependent anemia using 1.5T and 3T MRI scanner. | up to 1 week after the end of chelation therapy

SECONDARY OUTCOMES:
To calculate the T2* values in the pancreas, myocardium and pituitary gland in patients with transfusion-dependent anemia on the 3T scanner. | point1: Initially, after one month of chelation therapy; point 2: every week during 1 month for the stability checking point 3: ut to 1 week at the end of the study
To develop a control method for iron assessment using aqueous solutions of iron nanoparticles by calculating T2* values on 3T and 1,5T scanners. | point1: Initially, after one month of chelation therapy; point 2: every week during 1 month for the stability checking point 3: ut to 1 week at the end of the study
Draw up T2* values recalculating tables for a 3T scanner based on the distribution of T2* values for a 1.5T scanner in pancreas, myocardium, and pituitary gland in patients with transfusion-dependent anemia. | point1: Initially, after one month of chelation therapy; point 2: every week during 1 month for the stability checking point 3: ut to 1 week at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Galina f Tereshchenko, PhD, Study Director — Chief radiology department
Locations (1):
- Dmitry Rogachev National Medical Research Center Of Pediatric Hematology, Oncology and Immunology, Moscow, Samory-Mashela,1, Russia

IPD SHARING:
Plan to Share IPD: No